CLINICAL TRIAL: NCT02048241
Title: Intuniv vs Placebo in the Treatment of Childhood Intermittent Explosive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Stephen Donovan, Clinical Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #6068
Record Dates: First submitted 2012-12-13; First posted 2014-01-29 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Intermittent Explosive Disorder; Childhood Aggression; Oppositional Defiant Disorder; Attention Deficit Disorder
Keywords: childhood; temper; explosive; aggression; tantrums; oppositional; defiant; conduct; disruptive; emotional dysregulation; special education
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders; Oppositional Defiant Disorder; Attention Deficit Disorder with Hyperactivity; Aggression; Behavior | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo plus Parent Management Training (Other): Pills matching Intuniv Tablets without active medication combined with weekly Parent Management Training
  Interventions: Behavioral: Parent Management Training; Other: Placebo
- Intuniv plus Parent Management Training (Experimental): Administration of Intuniv in increasing doses from 1 mg to 2 mgs to 3 mgs to 4 mgs as tolerated over a period of 4-6 weeks, combined with weekly Parent Management Training
  Interventions: Behavioral: Parent Management Training; Drug: Intuniv

INTERVENTIONS:
Behavioral: Parent Management Training — This is a psychological treatment that focuses on decreasing tantrums and outbursts by reducing the ability of the tantrum to coerce parents into giving in to the demand that precipitated the tantrum.
  Other Names: PMT
Other: Placebo — Weekly dispensation of pills matching Intuniv but without the active medication
  Arms: Placebo plus Parent Management Training
Drug: Intuniv — Weekly administration of medication in doses as per protocol
  Other Names: Extended release Guanfacine
  Arms: Intuniv plus Parent Management Training

SUMMARY:
Children with explosive aggression are often rejected by their peers, placed in special classroom, and contribute to family discord. When psychotherapy and family therapy is unsuccessful, medications are often used. Current medications are stimulants (e.g. methylphenidate, dextroamphetamine), anticonvulsants (e.g. Divalproex) and antipsychotics (olanzapine, risperidone). At this time, the available medications are of limited usefulness, either because they do not always work or because they have side effects such as weight gain or insomnia. There is a clear need for new medications to treat explosive aggression when psychotherapy is unsuccessful.

The hypothesis of this study is the medication Intuniv when combined with psychotherapy will be more helpful to children with explosive aggression than placebo combined with psychotherapy. Intuniv is a long acting form of guanfacine, a medication approved by the FDA for treatment of Attention Deficit Hyperactivity Disorder. Intuniv is not a stimulant, nor is it an anticonvulsant, nor is it an antipsychotic.

The children in this study will be between the ages of 6 and 12 and meet Diagnostic and Statistical Manual of Psychiatry Fourth Edition, Text Revision (DSM-IV-TR) criteria for Intermittent Explosive Disorder.

DETAILED DESCRIPTION:
Aggressive children are often alienated from parents, separated from peers, placed in special education and segregated with other aggressive children. While predatory (i.e. planned, goal directed, reward driven) aggression is not responsive to pharmacologic treatment, non predatory (impulsive, paranoid, irritable) aggression (DSM-IV-TR "Intermittent Explosive Disorder") often is. Intermittent Explosive Disorder is characterized by discrete episodes of failure to resist aggressive impulses resulting in serious assaults or destruction of property. In children, due to their limited ability to damage or hurt others, the seriousness of the aggressive impulses are indicated by (a) the frequency and severity of tantrums (b) the fact that the severity is out of proportion to the provocation, and (c) the intent to damage and hurt is present and (d) this pattern of events causes impairment.

The level of aggression being studied is equivalent to that in moderate to severe Oppositional Defiant Disorder with the severity due to the tantrums rather than passive aggression (Modified Overt Aggression Score between 15-50). For 20 years a blood pressure medication, guanfacine (Tenex), has also been used for impulse control (e.g. in Attention Deficit Disorder, in Tourette's Syndrome) and to calm the sympathetic nervous system when it is hyper-aroused (e.g. in opiate and nicotine withdrawal]. Both impulsivity and hyper arousal can also promote intermittent explosive aggression. If guanfacine treats impulsivity and hyper arousal, it is logical to ask if guanfacine can treat intermittent explosive aggression.

Shire Pharmaceuticals modified the guanfacine molecule to create a long acting preparation (Intuniv) that the FDA recently judged safe and effective for Attention Deficit Hyperactivity Disorder (ADHD) in children ages 6-17. Secondary analysis of data from the pivotal studies that led to this indication revealed that in ADHD children, Intuniv also reduced oppositional-defiant symptoms. Better impulse control (these were all ADHD children) and/or decreased sympathetic arousal (common to all intermittent explosive aggression) are plausible explanations.

This Investigator Sponsor Protocol (ISP) seeks to replicate prospectively the anti-aggression finding. Since Intuniv could benefit non-ADHD aggressive children, any child with mild to moderate Intermittent Explosive Disorder is eligible. Anti-psychotic and anti-convulsant medications (current treatments for Intermittent Explosive Disorder) have serious side effects (weight gain, metabolic syndrome) and are not always effective. Intuniv is neither a stimulant, nor an antipsychotic, nor an anticonvulsant. Intuniv is not FDA approved for treatment of Intermittent Explosive Disorder.

In addition to medication or placebo, all children will receive a modified form of Parent Management Training, the standard psychotherapy for oppositional symptoms, administered by a child psychiatrist. It addresses the coercive reciprocal social interactions that characterize microenvironment of oppositional children.

Fifty children, ages 6-12 with Intermittent Explosive Disorder will be randomly assigned to eight weeks of double blind Intuniv plus Parent Management Training or placebo Parent Management Training. Titrated over four weeks to a maximum dose of 4 mgs or .09-.12 mgs/kg/day, they will be maintained on that dose for four weeks. At the end of treatment, the treating physician will break the blind and offer open label treatment for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-12
2. Meets DSM-IV TR Criteria for Intermittent Explosive Disorder

   1. several discreet episodes of failure to resist aggressive impulses that result in serious assaultive acts or destruction of property
   2. the degree of aggressiveness is grossly out of proportion to any precipitating psychosocial stressors
   3. the aggressive episode is not better accounted for by another mental disorder
   4. duration of at least six months
   5. impairment in home, peer relations and / or school
3. Modified Overt Aggression Scale (MOAS) score > 15
4. Parent and child willing to consent to study
5. Inadequate response to psycho-social interventions (including school interventions)
6. Medically healthy with

   1. weight > 55 lb (25 kg)
   2. body mass index < 35
   3. normal blood pressure as defined by National Heart Lung and Blood Institute (below 95th percentile for age height and weight)
   4. normal response to orthostatic changes (no persistent fall in systolic/diastolic BP > 20/10 mm Hg within 3 minutes of assuming the upright position)
   5. normal electrocardiogram
   6. normal vital signs
   7. no history of intolerance of guanfacine.
7. If on another medication, willingness to discontinue if medication is judged ineffective after adequate trial or to remain on a constant optimized dose if it is partially effective

Exclusion Criteria:

1. Current Treatment with another alpha 2 blocker e.g. clonidine
2. Puberty
3. Meets criteria for Pervasive Developmental Disorder or Childhood schizophrenia
4. MOAS score > 50
5. weight < 55 lb or body mass index > 35
6. hypertension (Blood Pressure above 95th percentile for age height and weight)
7. Chronic hypotension (Blood Pressure at or below 5th percentile for age height and weight)
8. Orthostatic Hypotension fall in systolic/diastolic BP > 20/10 mm Hg within 3 minutes of assuming the upright position
9. QTc interval of > 440 milliseconds; Bradycardia; heart block diagnosed
10. history of seizure during the past 2 years (exclusive of febrile seizures)
11. Patients who had taken an investigational drug within 28 days
12. Intelligence Quotient < 70
13. Physical exam, EKG or laboratory results with any other significant abnormalities until reviewed by medicine.
14. Active suicidal or homicidal ideation or history of suicide attempts
15. Unequivocal manic or hypomanic Episode
16. Patients who meet criteria for Major Depression in pre-puberty will not be eligible for this study.
17. Axis I disorders that are current, severe and uncontrolled. Children with moderate Axis I pathology will be evaluated on a case by case basis and excluded if the other diagnosis is not ADHD but could still be the cause of the temper dyscontrol and the treatment is judged substandard.
18. Any other history of cardiovascular dysfunction
19. Positive Urine Toxicology
20. Children who have experienced prior adverse effects (physical or psychological) to either Tenex or clonidine
21. Any child who previously received Tenex and either did not tolerate it, or failed to respond to an adequate trial

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Donovan, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: Columbia University Clinical Trials link — http://sklad.cumc.columbia.edu/psychiatry/clinical_trials/View_Trial.php?ID=376&type=simple

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Plus Parent Management Training | Intuniv Plus Parent Management Training
Started | 5 | 6
Completed | 5 | 5
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Parent Management Training | Intuniv Plus Parent Management Training | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 6 | 11
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 5 | 5 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 1 | 3
  African American | 1 | 2 | 3
  Hispanic | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Were Responders
Description: Overall response to treatment is defined as at least a 70% decline in both the Modified Overt Aggression Scale (MOAS) score and the Symptom Checklist-6 (SCL-6) from randomization to end of study. The MOAS measures the severity of explosive overt aggression. The score can range from 0 (no overt aggressive) and it has no theoretical upper limit (incidents could be too many to count). The higher the score, the more serious the aggression; the lower the score, the less serious the aggression. Response to treatment is defined as a 70% or more reduction in the MOAS at the end of the study. The SCL-6 uses 6 subscale items from the larger SCL that measure hostility or irritability on a scale of 1 (not at all) - 5 (definitely). The raw score ranges from 6 (no irritability) to 30 (severe irritability). The lower the score is, the better the outcome. The % decline vary from 0%-100%. A 70% or more decline in the SCL-6 score at the end of study is a response.
Time Frame: up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Plus Parent Management Training | Intuniv Plus Parent Management Training
Number analyzed (Participants) | 5 | 6
Participants | 0 | 5

ADVERSE EVENTS:
Arm/Group | Placebo Plus Parent Management Training | Intuniv Plus Parent Management Training
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 2/5 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Plus Parent Management Training (N=5) | Intuniv Plus Parent Management Training (N=6)
Fatigue (General disorders) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes